CLINICAL TRIAL: NCT00540306
Title: Monitoring Functional Variation in the Breast During Menstrual Cycle by Using Diffuse Optical Spectroscopy
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bruce Tromberg,Ph.D.,Director, Beckman Laser Institute and Medical Clinic and Professor, Departments of Biomedical Engineering and Surgery, University of California, Irvine
Other Study IDs: 20054760
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Accessory; Breast Tissue
Keywords: breast tissue

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnostic Tool: Changes in physiological and optical properties in healthy pre-menopausal breast tissue during the menstrual cycle using Diffuse Optical Spectroscopy
  Interventions: Device: Diffuse Optical Spectroscopy

INTERVENTIONS:
Device: Diffuse Optical Spectroscopy — Changes in physiological and optical properties in healthy pre-menopausal breast tissue during the menstrual cycle using Diffuse Optical Spectroscopy
  Other Names: Diffuse Optical Spectroscopy Imaging

SUMMARY:
The purpose of this study is to do determine the changes in physiological and optical properties in healthy pre-menopausal breast tissue during the menstrual cycle using Diffuse Optical Spectroscopy. The Researcher can determine 1) how large variations in breast tissue components are 2) how predictable and repeatable these variations are 3) the effects of endogenous hormones on breast tissue physiology.

DETAILED DESCRIPTION:
Variations in breast physiology due to hormonal fluctuations during the menstrual cycle can correlate to quantitative changes in Diffuse Optical Spectroscopy functional parameters such as hemoglobin, lipid and water concentration and tissue scattering. Diffuse Optical Spectroscopy imaging can show increase blood flow in breast tissue after ovulation with a concomitant increase in mitotic activity, changes in hemoglobin concentration and in tissue scattering. Increases in fibroglandular breast tissue after ovulation have also been observed. Diffuse Optical Spectroscopy imaging can determine after time of ovulation has been detected during the two months of self-monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Pre-Menopausal female 18 years of age or older with normal breast tissue
* Undergoes regular menstrual cycle cycles that do not vary by more than 5 days

Exclusion Criteria:

* Peri-Menopausal and Post-Menopausal
* Subjects taking oral contraceptives or any birth control medications in the past six months
* Diagnosed with breast cancer or cancer survivor,a history of breast surgery
* Subjects taking light sensitive drugs for photodynamic therapy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primary care clinic, community sample
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2006-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Breast Tissue Physiology | 4 weeks
  Changes in physiological and optical properties in healthy pre-menopausal breast tissue during the menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Bruce J Tromberg, Ph.D, Principal Investigator — Beckman Laser Institute University of California Irvine
Locations (1):
- Beckman Laser Institute University of California Irvine, Irvine, California, United States